CLINICAL TRIAL: NCT07302815
Title: Preemptive Intravenous Micro-dose Dexmedetomidine to Prevent Emergence Agitation in Adult Patients Undergoing Septoplasty Surgeries: A Randomized Placebo Controlled Study
Brief Title: Preemptive Intravenous Micro-dose Dexmedetomidine to Prevent Emergence Agitation in Adult Patients Undergoing Septoplasty Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Salah Salem, lecturer of anesthesia, surgical intensive care and pain management, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR131061/11/25
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Emergence Agitation
Keywords: Emergence agitation; septoplasty surgeries; micro-dose Dexmedetomidine
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Experimental): 60 patients will receive preoperative micro dose of dexmedetomidine (0.3 µg /kg) in 50 ml 0.9% saline slow infusion over 10 minutes, 15 minutes before surgery.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): 60 patients will receive preoperative micro dose of dexmedetomidine (0.3 µg /kg) in 50 ml 0.9% saline slow infusion over 10 minutes, 15 minutes before surgery.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — micro dose of dexmedetomidine (0.3 µg /kg) in 50 ml 0.9% saline slow infusion over 10 minutes, 15 minutes before surgery.
  Arms: Dexmedetomidine group
Drug: Saline — 50 ml 0.9% saline slow infusion over 10 minutes, 15 minutes before surgery.
  Arms: Control group

SUMMARY:
This prospective randomized controlled study will be conducted to evaluate the effect of preoperative single, micro-dose of dexmedetomidine (0.3μg/kg) on the incidence and severity of EA in adults undergoing Septoplasty surgeries

DETAILED DESCRIPTION:
Emergence agitation (EA) is characterised by confusion, restlessness or aggressive behaviour during recovery from general anaesthesia. EA is more common following ear, nose, & throat (ENT) surgery. The exact cause and pathophysiology of EA are unknown, although risk factors include preschool age, preoperative anxiety, postoperative pain, nausea, vomiting, otolaryngology operations, and the use of inhalational anesthetics particularly sevoflurane. EA might cause injury, accidental removal of intravenous cannulation, self-extubation, post-operative wound bleeding and increase the nursing requirements in the post-anesthesia care unit (PACU). There are limited studies concerning adult EA, and although its prevalence is less than child EA, it carries more risk of injury due to serious uncontrolled behaviors. Intravenous (IV) anesthetics, sedatives and opioids are the most frequently utilized medications to manage EA, with variable success rates and significant potential to delay recovery and cause undesirable side-effects. Dexmedetomidine is a highly selective α2 agonist which produces sedation and anxiolysis through reduction in sympathetic central nervous system activity. It has a major advantage over other sedatives; it is associated with minimal respiratory depression. According to a recent meta-analysis, intraoperative administration of dexmedetomidine decreases postoperative pain and the incidence of EA in adults. Considering the short length of corrective nasal reduction surgery (CR), an intraoperative infusion of dexmedetomidine as an anesthetic adjuvant may prolong the anesthesia and recovery time. Low dose infusion of dexmedetomidine (0.2 µg /kg/h) has been reported to reduce incidence of EA and opioid consumption effectively in elderly patients undergoing cancer surgeries under GA. Previous studies have shown that a single dose of dexmedetomidine, not as a premedication, is also effective in reducing EA and facilitating smooth extubation after pediatric adenotonsillectomy. Also recent study reported the efficacy of pre-operative dexmedetomidine administration (1 μg/kg) in preventing EA in adults undergoing CR of a nasal bone fracture. Up till now no clinical studies investigated the efficacy of single pre-operative micro dose of dexmedetomidine in prevention of EA, so in this clinical study we hypothesize that preoperative micro dose of dexmedetomidine may be beneficial in mitigation of EA in short timed Septoplasty surgeries safely and without prolongation of recovery time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both gender aged 18 to 60 years with American Society of Anesthesiologists (ASA) Physical Status I or II, who were scheduled for septoplasty surgery under general anesthesia.

Exclusion Criteria:

* Patients declined to participate in the trial.
* History or clinical evidence of chronic obstructive pulmonary disease.
* History of renal or hepatic dysfunction, sleep apnea syndrome.
* Cognitive dysfunction or psychiatric disorder.
* Patients receiving beta blocker.
* Patients with anticipated difficult airway.
* Patients with electro cardiac abnormalities.
* Emergency surgeries.
* Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of emergence agitation | incidence of emergence agitation will be assessed by Aono's Four-point Scale (AFPS) after extubation, at PACU arrival, every 5 minutes for the first 15 minutes then every 15 minutes for the first hour after surgery.
  using Aono's Four-Point Scale (Aono Scale) which is a simple and widely used tool to assess emergence agitation (EA). It categorizes agitation during emergence from anesthesia into four levels.
  1. calm_ Patient is quiet and not agitated.
  2. Not calm but can be easily consoled _ Slight restlessness but settles with verbal reassurance or mild physical comfort.
  3. Moderately agitated _ Patient is crying or difficult to console but not combative.
  4. Severely agitated _Patient is thrashing, inconsolable, or combative, and poses risk of injury to self or staff.
  Scores 3-4 indicate clinically relevant emergence agitation.

SECONDARY OUTCOMES:
severity of emergence agitation | severity of EA will be assessed by Aono's Four-point Scale (AFPS) after extubation, at PACU arrival, every 5 minutes for the first 15 minutes then every 15 minutes for the first hour after surgery.
  Aono's Scale grades the intensity of a patient's agitation during emergence from anesthesia (3) Moderately agitated - Patient is crying or difficult to console but not combative.
  (4) Severely agitated - Patient is thrashing, inconsolable, or combative, and poses risk of injury to self or staff.
extubation time | Extubation time is the duration between the cessation of anesthetic agents and removal of endotracheal tube (ETT).
  Extubation time is the duration between the cessation of anesthetic agents and removal of endotracheal tube (ETT).
Length of stay in the post anesthetic care unit (PACU). | time from the moment they arrive after surgery until they meet discharge criteria and are officially transferred to the ward
  Total time a patient spends in the PACU from the moment they arrive after surgery until they meet discharge criteria and are officially transferred to the ward
Intraoperative opioid consumption | from induction of anesthesia until completion of surgery
  Total amount of opioid medications administered to a patient during the entire surgical procedure, from induction of anesthesia until completion of surgery
Post operative numerical rating scale score (NRS) | - NRS score is measured at PACU arrival and every 15 minutes for 1 hour after surgery
  The Numerical Rating Scale (NRS) is a validated tool used to assess a patient's pain intensity by having them assign a number to their pain on a 0-10 scale.
  On a scale from 0 to 10, where 0 means no pain and 10 is the worst pain imaginable

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: The data will be available upon a reasonable request from the corresponding author after the end of the study for one year
Access Criteria: The data will be available upon a reasonable request from the corresponding author

REFERENCES:
- [Background] Kim JC, Kim J, Kwak H, Ahn SW. Premedication with dexmedetomidine to reduce emergence agitation: a randomized controlled trial. BMC Anesthesiol. 2019 Aug 7;19(1):144. doi: 10.1186/s12871-019-0816-5. PMID 31391001
- [Background] Guler G, Akin A, Tosun Z, Ors S, Esmaoglu A, Boyaci A. Single-dose dexmedetomidine reduces agitation and provides smooth extubation after pediatric adenotonsillectomy. Paediatr Anaesth. 2005 Sep;15(9):762-6. doi: 10.1111/j.1460-9592.2004.01541.x. PMID 16101707
- [Background] Lee HS, Yoon HY, Jin HJ, Hwang SH. Can Dexmedetomidine Influence Recovery Profiles from General Anesthesia in Nasal Surgery? Otolaryngol Head Neck Surg. 2018 Jan;158(1):43-53. doi: 10.1177/0194599817733735. Epub 2017 Sep 26. PMID 28949804
- [Background] Abdelaziz TSA, Mohammed Elsayed HE, Kamal Eldin DM, Ibrahim IM. "The effect of intramuscular dexmedetomidine versus oral gabapentin premedication on the emergence agitation after rhinoplasty". A prospective, randomized, double-blind controlled trial. BMC Anesthesiol. 2025 Jan 31;25(1):50. doi: 10.1186/s12871-025-02914-5. PMID 39891093
- [Background] Zhu W, Sun J, He J, Zhang W, Shi M. A Randomized Controlled Study of Caudal Dexmedetomidine for the Prevention of Postoperative Agitation in Children Undergoing Urethroplasty. Front Pediatr. 2021 Sep 29;9:658047. doi: 10.3389/fped.2021.658047. eCollection 2021. PMID 34660472
- [Background] Al Mutair A, Alabbasi Y, Alshammari B, Alrasheeday AM, Alharbi HF, Aleid AM. A Meta-Analysis of the Impact of Intranasal Dexmedetomidine on Emergence Delirium and Agitation in Children and Adolescents Undergoing Tonsillectomy and/or Adenoidectomy. J Clin Med. 2025 Feb 26;14(5):1586. doi: 10.3390/jcm14051586. PMID 40095538
- [Background] Cole JW, Murray DJ, McAllister JD, Hirshberg GE. Emergence behaviour in children: defining the incidence of excitement and agitation following anaesthesia. Paediatr Anaesth. 2002 Jun;12(5):442-7. doi: 10.1046/j.1460-9592.2002.00868.x. PMID 12060332
- [Background] Yu D, Chai W, Sun X, Yao L. Emergence agitation in adults: risk factors in 2,000 patients. Can J Anaesth. 2010 Sep;57(9):843-8. doi: 10.1007/s12630-010-9338-9. Epub 2010 Jun 5. PMID 20526708
- [Background] Tolly B, Waly A, Peterson G, Erbes CR, Prielipp RC, Apostolidou I. Adult Emergence Agitation: A Veteran-Focused Narrative Review. Anesth Analg. 2021 Feb 1;132(2):353-364. doi: 10.1213/ANE.0000000000005211. PMID 33177329